Improvement of perimenstrual acne with clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel

PI: Anjali Vekaria NCT03122457

Document Date: July 22, 2015

| M |
|--------|
| ////// |
| Mount |
| Sinai |

| Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate |
|---|---|
| | and benzoyl peroxide 1.2%/3.75% combination gel |
| Principal Investigator | Anjali Shroff, MD |
| Name/Contact Info: | |
| Primary Contact | Matthew Gagliotti +1 212.241.3288 |
| Name/Contact Info | |
| Date Revised: | 22 July 2015 |
| Study Number: | HSM #15-00563 |

## **MSSM Protocol Template HRP-503**

- Note that, depending on the nature of your research, certain questions, directions, or entire sections below may not be applicable. Provide information if and when applicable, and in cases where an entire section is not applicable, indicate this by marking the section "N/A". Do not delete any sections.
- For any items below that are already described in the sponsor's protocol, the investigator's protocol, the
  grant application, or other source documents, you may simply reference the title and page numbers of
  these documents in the sections below, rather than cutting and pasting into this document. Do not refer to
  the Sample Consent document, or information on the application form in this document.
- Keep an electronic copy of this version of the document. You will need to modify this copy when making changes.

### **Brief Summary of Research (250-400 words):**

We plan to enroll a total of 40 subjects with perimenstrual acne. Eligible women will be over the age of 18 and not on any current therapy. They will first arrive for a screening visit, where they will be given questionnaires on acne quality of life (acne QOL) and subjective assessments as well as flare ups (as used in the study by Geller et al). Their skin will be assessed for inflammatory and non-inflammatory acne vulgaris. The Baseline visit (day 1) will be scheduled for one week prior to the day of their menses (as studies indicate that most women have their acne flare during this time). We will perform a zit count (counting papules, pustules, and comedones) and global assessment, and the patient will be instructed to record their menses (which they will do for the duration of the study). They will then return in 2 weeks, at day 15, and they will be reassessed. They will be dispensed the investigational product and instructed on its daily use. They will continue to return every 14 days to have their skin assessed until their final visit on day 99, one week after their 3<sup>rd</sup> menses on treatment (4<sup>th</sup> menses on study). The duration of the study per patient is approximately 4 months, and we anticipate an enrollment period of 12 months.

## 1) Objectives:

In this study, we will look at the effectiveness of clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel for perimenstrual acne. The gel is the first and only FDA-approved fixed combination of 1.2% clindamycin phosphate and 3.75% benzoyl peroxide medication, and has been proven effective in the treatment of comedonal (non-inflammatory) and inflammatory acne when used once daily. We hope to demonstrate its effectives as a single agent in treating perimenstrual acne.

| M |
|-------|
| /// |
| Mount |
| Sinai |

| Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate |
|---|---|
| | and benzoyl peroxide 1.2%/3.75% combination gel |
| Principal Investigator | Anjali Shroff, MD |
| Name/Contact Info: | |
| Primary Contact | Matthew Gagliotti +1 212.241.3288 |
| Name/Contact Info | |
| Date Revised: | 22 July 2015 |
| Study Number: | HSM #15-00563 |

### 2) Background

Acne is an extremely common dermatologic problem, affecting over 17 million individuals in the United States. While it is typically thought of as a disorder affecting adolescents, many individuals continue to have acne or first develop acne in adulthood. Among those over the age of 20, acne is more commonly seen in females than in males, and in this female population it is often perceived as perimenstrual. One study performed at Mount Sinai demonstrated that of 105 adult women with acne, 65% felt that their acne worsened perimenstrually.

Due to the significant role of androgens in the development of perimenstrual acne, hormonal therapy with oral contraceptive pills or spironolactone has long been a mainstay of treatment. Yet for many women, these therapies are problematic due to their side effects, stigma, or pill burden. Topical treatments are often used as well; however, at present no topical therapy has been demonstrated to be more effective in women with this type of hormonal acne.

### 3) Setting of the Human Research

Subjects will attend their study visits in the outpatient offices at the FPA, 5<sup>th</sup> floor, Department of Dermatology.

## 4) Resources Available to Conduct the Human Research

In the past we never have had any difficulty recruiting potential study patients, particularly for studies that focus upon acne. We will mostly rely on our database of potential subjects who have requested to be contacted for future studies. In addition, we have a very active referral base from the in-house residents, and affiliated attendings. Thus, the recruitment of the 40 required subjects for this study should not be difficult, and our timelines should be met with ease.

Our staff is very well versed and experienced in conducting clinical trials. For further information, please locate the PI and sub-investigators' Curriculum Vitae.

All Persons assisting with the trial have copies of the protocol, and knowledge of the study drugs involved in the trial.

| M |
|-------|
| //// |
| Mount |
| Sinai |

| Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel |
|---|---|
| Principal Investigator | Anjali Shroff, MD |
| Name/Contact Info: | |
| Primary Contact | Matthew Gagliotti +1 212.241.3288 |
| Name/Contact Info | |
| Date Revised: | 22 July 2015 |
| Study Number: | HSM #15-00563 |

## 5) Study Design

### a) Recruitment Methods

Potential subjects will come from our database of patients who have requested to be contacted for future studies, and they will be referred by in-house residents and affiliated attendings. In addition, IRB approved advertisements will be used.

### b) Inclusion and Exclusion Criteria

Please see page 3 of the protocol under sections, « Inclusion Criteria » and « Exclusion Criteria ».

## c) Number of Subjects

Forty people are expected to take part in this clinical trial. This is a single-center study, which will only be conducted at Mount Sinai.

### d) Study Timelines

The study duration for each subject will be 99 days. We anticipate beginning enrollment in August 2015, and expect to complete the enrollment of all 40 subjects by June 2016. Therefore, the last patient visit should occur in October 2016. We will require another 2-3 months to complete all data analyses. We expect to complete the entire study, including analyses by January 2017.

## e) Study Endpoints

Please see page 7 of the protocol under section, « Efficacy Endpoints ».

## f) Procedures Involved in the Human Research

Please see page 4 of the protocol under section, « Study Methodology ».

The subject's medical history and any concomitant or past medications/ therapies will be collected from the patient via his/her recollection. No chart review will be performed.

Provided subject consent, photographs will be taken at each visit. Digital photographs of the subject will be taken to record the location and extent of acne. Photo consent is not mandatory for participation in this study. If the photos are used in publications, the eyes will be blackened out to protect the identity of the subjects.

Female subjects of childbearing potential must consent to a urine pregnancy test.

| N | A |
|-------------|---|
| Mou<br>Sina | |

| Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel |
|---|---|
| Principal Investigator<br>Name/Contact Info: | Anjali Shroff, MD |
| Primary Contact | Matthew Gagliotti +1 212.241.3288 |
| Name/Contact Info | |
| Date Revised: | 22 July 2015 |
| Study Number: | HSM #15-00563 |

### g) Specimen Banking

N/A

## h) Data Management and Confidentiality

All records, including photographs, identifying the subject will be kept confidential and, to the extent permitted by the applicable laws and/or regulations, will not be made publicly available. Subject names will not be supplied to the sponsor. Only the subject number will be recorded in the CRF, and if the subject name appears on any other document, it must be obliterated before a copy of the document is supplied to the sponsor. Study findings stored on a password protected computer will be encrypted and stored in accordance with local data protection laws. Only the PI, sub-investigators, and main study coordinator (back-up coordinator, if applicable) will have access to the data that is collected. As part of the informed consent process, the subjects will be informed in writing that representatives of the sponsor, IRB, or regulator authorities may inspect their medical records to verify the information collected, and that all personal information made available for inspection will be handled in strictest confidence and in accordance with local data protection laws. If the results of the study are published, the subject's identity will remain confidential. Only the investigator will maintain a list to enable subjects to be identified.

## i) Provisions to Monitor the Data to Ensure the Safety of subjects

This information is only required when Human Research involves more than Minimal risk to subjects.

**Part I** describes the safety monitoring activities that will be undertaken in during the study. This should be completed for all studies that require more than the basic minimum DSMP. **Part II** describes Data and Safety Monitoring Committees or Boards and should be completed when one is needed for the DSMP

### Part I: Elements of a Data and Safety Monitoring Plan

1. List the name(s) of the individual(s) at MSSM who will be responsible for data and safety monitoring of this study. For each individual, indicate their role, name, title, and department information. The Principal Investigator may be the only monitor of a study. If the qualifications of an individual to serve as a monitor are not contained in the PPHS application, they must be added to the DSMP either as a narrative description or as a CV.

| | Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel |
|---|---|---|
| Mount<br>Sinai | Principal Investigator Name/Contact Info: | Anjali Shroff, MD |
| | Primary Contact Name/Contact Info | Matthew Gagliotti +1 212.241.3288 |
| Sinai | Date Revised: | 22 July 2015 |
| | Study Number: | HSM #15-00563 |

### **MSSM Principal Monitor:**

Indicate whether this person is the PI, a Team Member, or is Independent: Last Name:

Goldenberg
First Name: Gary

Academic Title: Assistant Professor

Department: Dermatology

Mailing Address: New York, NY 10029 USA

Phone: +1 212.241.3288

Fax: N/A

Email: gary.goldenberg@mounsinai.org

#### **MSSM** Additional Monitor:

Indicate whether this person is the PI, a Team Member, or is Independent:

Last Name: Shroff First Name: Anjali

Academic Title: Dermatopharmacology research fellow

Department: Dermatology

Mailing Address: New York, NY 10029 USA

*Phone:* +1 212.241.3288

Fax: N/A

Email: Anjali.shroff@mssm.edu

- 1. The principal monitor is the most experienced investigator on this study. Please refer to respective curriculum vitae for further information.
- 2. Please see protocol page 6, under «Safety Evaluations». Early termination subjects will be asked for one last follow-up to track their final progress. Safety and AEs will be assessed at each visit.
- 3. The sum of safety data will be analyzed upon stud completion, as this is a short-term study. Any significant safety data will be reported to the sponsor.
- 4. With regards to subject withdrawal or discontinuation, subjects may choose to withdraw from the study or be withdrawn by the investigator at any time without prejudice to their future medical care. Any subject who does not comply with the inclusion/exclusion criteria may be withdrawn from further participation in the study. Any subject who receives study product and discontinues prematurely from the study should return to the stud center for an End of Study Visit.
- **5.** N/A
- **6.** Adverse events will be recorded on the source for each patient during each study visit. A local skin reaction grading system will be used for recording the severity of adverse events.
- 7. Each sub-investigator will sign/initial the source sheet for each visit after ensuring that all the required data is recorded accurately.
- **8.** Should a temporary or permanent suspension of your stud occur, in addition to the PPHS, we will report the occurrence to the IRB.

| | Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel |
|---|---|---|
| | Principal Investigator<br>Name/Contact Info: | Anjali Shroff, MD |
| Mount<br>Sinai | Primary Contact<br>Name/Contact Info | Matthew Gagliotti +1 212.241.3288 |
| Sina | Date Revised: | 22 July 2015 |
| | Study Number: | HSM #15-00563 |

## j) Withdrawal of Subjects

Any subject who discontinues, for any reason, will be encouraged to return for a final visit in order to collect safety data (disease assessment (PGA); photographs; adverse event assessment; concomitant medication documentation).

### 6) Risks to Subjects

Risks from the study drug commonly include: burning sensations, contact dermatitis, pruritus, and rash in the treatment area. Additionally, although uncommon, systemic absorption of clindamycin (clindamycin being absorbed through your skin into your blood) has been reported following its topical use. Diarrhea, bloody diarrhea, and colitis have been reported with the use of topical and systemic clindamycin. If significant diarrhea occurs, the study drug should be discontinued.

Allergic reactions, including anaphylaxis, have also rarely been reported.

Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.

If you are or become pregnant, this research may hurt your baby or your pregnancy in ways that are unknown. The unknown risks might be minor or might be major (death). You should not become pregnant while you are on this research study.

In addition to these risks, this research may hurt you in ways that are not known. The unknown risks might be minor or might be major (death).

## 7) Provisions for Research Related Injury

If a subject is injured or made sick from taking part in this research study, medical care will be provided. Generally, this medical care will be billed to the subject and/or the subject's health care insurance. In some cases, the costs of this care may be paid by someone else. In the event of injury, contact the Principal Investigator.

If the subject follows the directions of the study doctor and staff and the subject is physically injured because of a properly given drug, or procedures necessary for this study, the sponsor will pay the medical expenses for the treatment of that injury which are not covered by the subject's medical insurance, by a government program, or by any other third party.

## 8) Potential Benefits to Subjects

Since the study drug being used commonly treats acne, there is a reasonable chance that this study may benefit the subjects. The possible benefit is that the subjects' acne may clear.

## 9) Provisions to Protect the Privacy Interests of Subjects

All results and data will be collected and analyzed within Mount Sinai. Patient documents will be stored in a secure place. Staff at Mount Sinai school of Medicine Dermatology Clinical Trials department has to undergo IRB and HIPAA training. Only the investigators,



| Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate |
|---|---|
| | and benzoyl peroxide 1.2%/3.75% combination gel |
| Principal Investigator | Anjali Shroff, MD |
| Name/Contact Info: | |
| Primary Contact | Matthew Gagliotti +1 212.241.3288 |
| Name/Contact Info | - |
| Date Revised: | 22 July 2015 |
| Study Number: | HSM #15-00563 |

sub-investigators and study coordinator will have access to this data. Patient photographs will be stored in a secure folder that only people listed in the study will have access to.

Only subjects who have given us permission to contact them for studies will be contacted. All conversations with subjects and potential subjects will be conducted in a private examination room with the subject. Family members will be allowed to remain in the room only if the subject allows it. If the subject must be contacted by phone, then the study staff will only speak to the subject, and if a message is required, no information regarding the subject's disease, treatment or the fact that he/she is involved in a study will be conveyed.

### 10) Economic Impact on Subjects

Patients will be compensated \$25 per study visit for transportation, excluding screening. The study medications will be of no cost to the subject.

## 11) Payment to Subjects

Subjects will be paid \$25 per study visits 1-8 totaling \$125. Since this is a short study, subjects will be paid upon completion.

Subjects who do not complete all study visits will be compensated for those which have been completed.

## 12) Consent Process

HRP-090 Informed Consent Process for Research will be followed.

The Consent will be obtained prior to any study procedures and administered by the Principal Investigator or delegates. The consent process will be performed either at the first visit to the study site (not necessarily the first stud visit as specified in the protocol) or should the subject prefer to take the consent home to read at leisure, at a subsequent visit. Consent will be obtained in a private, closed-door patient room which will not permit others to overhear the consent process. The Screening Visit will occur immediately after consent is obtained. No study procedures will be performed until written consent is provided.

If necessary, in cases where the subject does not speak/read English, a translator will be used and an IRB approved consent form in his/her native language will be used. If a potential subject requires a consent form in a specific language which cannot be obtained, that that subject will not be eligible to participate in this stud. The Screening Visit will occur immediately after consent is obtained. No study procedures will be performed until written consent is provided.

Subjects are required to provide their date of birth at the first visit. We use this information to document the subject's legal age. If we feel a date is questionable we ask for a photo ID. Should the subjects have a birthday that makes them under 18 years of age the will not be enrolled in this study.

| | Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel |
|---|---|---|
| Mount<br>Sinai | Principal Investigator<br>Name/Contact Info: | Anjali Shroff, MD |
| | Primary Contact<br>Name/Contact Info | Matthew Gagliotti +1 212.241.3288 |
| Diriu: | Date Revised: | 22 July 2015 |
| | Study Number: | HSM #15-00563 |

## 13) Process to Document Consent in Writing

This study will be using the standard PPHS consent template.

### 14) Vulnerable Populations

Indicate specifically whether you will include (target) or exclude each of the following populations:

| Include | Exclude | Vulnerable Population Type |
|---|---|---|
| | V | Adults unable to consent |
| | V | Individuals who are not yet adults (e.g. infants, infants, teenagers) |
| | V | Wards of the State (e.g. foster children) |
| | √ | Pregnant women |
| | V | Prisoners |

# 15) Multi-Site Human Research (Coordinating Center)

N/A

## 16) Community-Based Participatory Research

N/A

# 17) Sharing of Results with Subjects

It is a requirement that the study subject's involvement in this study be noted in his or her medical records. If the study subject's primary care physician is different from the study doctor for this study, the PCP may also be notified of the subject's involvement in this study.

Direct access to the study subject's records will be require by authorized representatives of the sponsor to check the information collected for the study. Medical records may also be reviewed and copies made by members of either the institutional review

| | Protocol Title: | Improvement of perimenstrual acne with clindamycin phosphate and benzoyl peroxide 1.2%/3.75% combination gel |
|---|---|---|
| Mount<br>Sinai | Principal Investigator | Anjali Shroff, MD |
| | Name/Contact Info: | |
| | Primary Contact | Matthew Gagliotti +1 212.241.3288 |
| | Name/Contact Info | |
| | Date Revised: | 22 July 2015 |
| | Study Number: | HSM #15-00563 |

board/independent ethics committee responsible for this study site, regulatory agencies in countries where approval for the investigational products may be sought and/or authorized representatives of the sponsor. These individuals will see the subject's name, other personal information such as date of birth and gender, and medical information, but should not disclose the subject's name to anyone else. However, because of the need for these parties to have access to medical information, absolute confidentiality cannot be guaranteed.

## 18) IRB Review History

N/A

### 19) Control of Drugs, Biologics, or Devices

Study drug is stored in a temperature-controlled, combination-locked room accessible only by clinical trials personnel. It will be dispensed to eligible subjects by PI-delegated study personnel.